CLINICAL TRIAL: NCT00934947
Title: The BURN HELP Trial: BURN Healing and AnaLgesia With Propranolol
Brief Title: Burn Healing and Analgesia With Propranolol
Acronym: BURN HELP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-0681
Record Dates: First submitted 2009-07-06; First posted 2009-07-08 (Estimated); Results first posted 2012-10-29 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-09

CONDITIONS: Burns; Pain
Keywords: Burns; Pain
MeSH Terms: conditions — Burns; Pain | interventions — Propranolol; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sugar pill (Placebo Comparator)
  Interventions: Drug: Placebo
- Propranolol, Propanolol ER (Experimental)
  Interventions: Drug: Propranolol; Drug: Propanolol

INTERVENTIONS:
Drug: Propranolol — 40 mg
  Other Names: Inderal; Innopran
  Arms: Propranolol, Propanolol ER
Drug: Placebo — sugar pill
  Other Names: Sugar pill
  Arms: Sugar pill
Drug: Propanolol — 120 mg twice per day
  Other Names: Inderal; Innopran
  Arms: Propranolol, Propanolol ER

SUMMARY:
The purpose of this study is to investigate the ability of propranolol to decrease pain and improve recovery in burn patients with a common genotype.

ELIGIBILITY:
Inclusion Criteria:

* Thermal burn
* Greater than or equal to 18 years of age
* Less than 60 years of age
* Able to speak and read English

Exclusion Criteria:

* Intubated
* Clinically unstable
* Other substantial comorbid injury (e.g. long bone fracture)
* Heart block greater than first degree (EKG)
* History of coronary artery disease
* History of congestive heart failure
* Asthma (within past 10 years, induced by a beta-blocker, or receiving current treatment)
* Pregnant
* Prisoner
* Psychotic, suicidal, or homicidal
* Diabetic
* Hepatic failure (acute or chronic)
* Renal failure (acute or chronic)
* History of hyperthyroidism unless taking synthroid or other thyroid hormone replacement
* Exceeds daily acceptable chronic opioid use prior to burn
* Interacting medication
* Received propranolol within the last 6 months
* Multiple severe allergic reactions
* On daily methylphenidate or similar stimulant medication
* Unwilling to use medically acceptable birth control (if childbearing potential)
* Breastfeeding
* Severe peripheral vascular disease or vasospastic disorder
* Bradycardia that in the opinion of the investigator would constitute too great a risk when considered in the context of the patient's medical comorbidities and health history
* Other criteria that in investigator's opinion makes participant poor candidate for the trial
* Cancer (except basal cell cancer)

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2009-07; Primary Completion 2011-02 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel McLean, MD, MPh, Principal Investigator — University of North Carolina, Department of Anesthesiology
Locations (4):
- United States (4):
  - Washington Hospital Center, Washington D.C., District of Columbia
  - North Carolina Jaycee Burn Center, Chapel Hill, North Carolina
  - Wake Forest University Baptist, Wake Forest, North Carolina
  - Crozer Chester Medical Center, Upland, Pennsylvania

REFERENCES:
- See also: NC Jaycee Burn Center — http://www.med.unc.edu/burn

RESULTS

PARTICIPANT FLOW:
Groups:
- Sugar Pill: Identical to active drug in sight, taste, and smell.
- Propranolol, Propanolol ER: Identical to sugar pill in sight, taste, and smell.
Period: Overall Study
Arm/Group | Sugar Pill | Propranolol, Propanolol ER
Started | 23 | 22
Completed | 23 | 20
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugar Pill | Propranolol, Propanolol ER | Total
Number analyzed (Participants) | 23 | 22 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 22 | 45
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (11) | 31 (9) | 32 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 19 | 15 | 34
Region of Enrollment [Number; unit: participants]
  United States | 23 | 22 | 45

OUTCOME MEASURES:

1. Primary Outcome: Overall Pain Trajectory Slopes
Description: Overall pain trajectory slopes by treatment group, where linear mixed modeling was used to combine pain measurements (waking, worst, and least pain) assessed on primary outcome days into an overall pain score. Pain was assessed using a 0-10 numeric rating scale (NRS). A lower score on the NRS indicated less pain and a higher score was indicative of worse pain.
Time Frame: Study days 5, 7, 10, 13, 17 and 19
Measure: Least Squares Mean (95% Confidence Interval); unit: Numeric Rating Scale Score Change/Day
Arm/Group | Sugar Pill | Propranolol, Propanolol ER
Number analyzed (Participants) | 23 | 20
Numeric Rating Scale Score Change/Day | -0.22 [-0.25 to -0.19] | -0.16 [-0.19 to -0.13]

2. Secondary Outcome: Sleep Quality
Description: Medical Outcomes Survey Sleep Quality Subscale. This is a 0-10 numeric rating scale in which patients rate their sleep quality. 0 represents poor sleep quality whereas 10 represents a restful night of sleep.
Time Frame: 6 weeks after injury timepoint was chosen for this analysis
Population: The number of participants who reported sleep quality at the 6 week time point are included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Propranolol: Individuals who were randomized to receive propranolol following an intention to treat analysis
- Placebo: Individuals enrolled in the study who received placebo
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 16 | 22
units on a scale | 6.75 (2.49) | 7.46 (2.02)
Statistical Analysis 1: Comparison: Propranolol vs Placebo; Test type: Superiority; p = .36, t-test, 2 sided

3. Secondary Outcome: Itch Symptoms
Description: Average itch intensity measured with a 0-10 numeric rating scale, 6 weeks was used as main outcome timepoint for itch symptom burden. 0 represents no itch symptoms and 10 represents the most severe itch symptoms.
Time Frame: Week 6 after injury was chosen as the main timepoint of interest
Population: The number of participants who reported itch at the 6 week time point are included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 16 | 22
units on a scale | 1.91 (1.81) | 2.61 (2.89)
Statistical Analysis 1: Comparison: Propranolol vs Placebo; Test type: Superiority; p = .32, t-test, 2 sided

4. Secondary Outcome: Anxiety Symptoms
Description: Anxiety severity via the State Trait Personality Inventory (STPI), range 10-40, 40 represents high anxiety.
Time Frame: 6 weeks after injury was chosen as the main timepoint of interest
Population: The number of patients represents the number of participants responding at 6 weeks after injury.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 15 | 22
units on scale | 15.27 (4.62) | 14.23 (3.87)
Statistical Analysis 1: Comparison: Propranolol vs Placebo; Test type: Superiority; p = .48, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Sugar Pill | Propranolol, Propanolol ER
Serious Adverse Events (participants affected / at risk) | 1/23 | 0/22
Other Adverse Events (participants affected / at risk) | 6/23 | 8/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugar Pill (N=23) | Propranolol, Propanolol ER (N=22)
Thrombisis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugar Pill (N=23) | Propranolol, Propanolol ER (N=22)
Nausea (Gastrointestinal disorders) | 6 (6) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No